CLINICAL TRIAL: NCT01556763
Title: A Double-Blind, Placebo-Controlled Randomized Study to Assess the Safety, Tolerability, and Pharmacokinetics of EVP-6124 in Participants With Schizophrenia on Stable Monotherapy With Selected Antipsychotics
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of EVP-6124 in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EVP-6124-005
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Central Nervous System Diseases
Keywords: Schizophrenia; Schizoaffective; CNS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Central Nervous System Diseases | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo was administered as one capsule per day for 21 days.
  Interventions: Drug: Placebo; Drug: Antipsychotic therapy
- EVP-6124 (1.0 mg/day) (Experimental): EVP-6124 was administered as one 1.0 mg capsule per day for 21 days.
  Interventions: Drug: EVP-6124 (1.0 mg/day); Drug: Antipsychotic therapy
- EVP-6124 (0.3 mg/day) (Experimental): EVP-6124 was administered as one 0.3 mg capsule per day for 21 days.
  Interventions: Drug: EVP-6124 (0.3 mg/day); Drug: Antipsychotic therapy

INTERVENTIONS:
Drug: EVP-6124 (0.3 mg/day) — EVP-6124 was administered as one 0.3 mg capsule per day for 21 days.
  Arms: EVP-6124 (0.3 mg/day)
Drug: EVP-6124 (1.0 mg/day) — EVP-6124 was administered as one 1.0 mg capsule per day for 21 days.
  Arms: EVP-6124 (1.0 mg/day)
Drug: Placebo — Matching placebo was administered as one capsule per day for 21 days.
  Arms: Placebo
Drug: Antipsychotic therapy — Concomitant therapy with antipsychotic medication (aripiprazole [10 to 30 mg/day], olanzapine [10 to 20 mg/day], paliperidone [3 to 12 mg/day], or risperidone [2 to 16 mg/day]), taken at the same time each day as the EVP-6124 dose. Patients must have been taking concomitant therapy for at least 2 weeks at a stable dose to be eligible for the study.

SUMMARY:
This study in patients with schizophrenia is designed to provide preliminary evidence of the safety, tolerability, and pharmacokinetics as well as the effects on cognitive function of 2 doses of EVP-6124 compared with placebo when given with the patient's usual antipsychotic medication.

DETAILED DESCRIPTION:
Study drug will be supplied as capsules and will be orally administered once daily for a total of 21 days. Eligible subjects will be admitted to an inpatient study unit on Day -6 (six days before the first dose of study drug is administered) and will remain confined to the inpatient study unit throughout the dosing phase. Safety assessments, PK sampling, and cognitive testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 55 years (both inclusive).
* Females must be surgically sterile, post-menopausal, or using reliable contraception and have negative pregnancy tests at screening and at Day -1.
* A clinical diagnosis of schizophrenia or schizoaffective disorder and prescribed a stable dose of aripiprazole (10 to 30 mg/day), olanzapine (10 to 20 mg/day), paliperidone (3 to 12 mg/day), or risperidone (2 to 16 mg/day) for a minimum of 2 weeks before initial screening.
* In good general health and expected to complete the clinical trial as designed.
* Body Mass Index (BMI) of 18 kg/m^2 to 38 kg/m^2 (both inclusive) at screening.
* Adequate hearing, vision, and language skills to perform the cognitive testing and other procedures specified in the protocol.
* Voluntarily provided informed consent and signed an informed consent form (ICF) indicating that the purpose of the study was explained, and was willing and able to adhere to the study regimen and study procedures described in the ICF, including all confinement requirements.
* Negative urine drug screen at screening and inpatient observation baseline period (Day -6), except for a short-acting benzodiazepine if prescribed for insomnia.
* Fluent in English (speaking, writing, and reading).

Exclusion Criteria:

* Female subject who was pregnant or breast-feeding.
* Any active clinically significant medical condition within 1 month (30 days) prior to screening.
* A history of substance (drug) dependence or substance or alcohol abuse within the 12 months before randomization as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV).
* A score of >5 on any item on the PANSS (Positive and Negative Syndrome Scale) Positive subscale at baseline during the inpatient observation period (Day -1).
* Any laboratory test abnormalities at screening indicating hepatic or renal dysfunction, or any other laboratory test abnormalities deemed by the investigator to be clinically significant.
* Any hematologic malignancy or solid tumor diagnosed within 3 years prior to study entry with the exception of localized skin cancer or carcinoma in situ of the cervix.
* Known to have had or was a carrier of HBsAg, HCV antibody, or had a positive result to the HIV-1 and/or HIV-2 antibodies.
* Uncooperative with or could not complete the study procedures.
* Received an investigational drug within 30 days before screening.
* Donated blood within 30 days before randomization on Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon H. Preskorn, M.D., Principal Investigator — Clinical Research Institute
Locations (1):
- Clinical Research Institute, Wichita, Kansas, United States

REFERENCES:
- [Derived] Preskorn SH, Gawryl M, Dgetluck N, Palfreyman M, Bauer LO, Hilt DC. Normalizing effects of EVP-6124, an alpha-7 nicotinic partial agonist, on event-related potentials and cognition: a proof of concept, randomized trial in patients with schizophrenia. J Psychiatr Pract. 2014 Jan;20(1):12-24. doi: 10.1097/01.pra.0000442935.15833.c5. PMID 24419307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Started | 4 | 9 | 8
Completed | 4 | 8 | 8
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day) | Total
Number analyzed (Participants) | 4 | 9 | 8 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 9 | 8 | 21
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.0 (11.6) | 43.1 (11.0) | 51.4 (6.9) | 45.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 6
  Male | 4 | 6 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 4 | 9 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Spontaneously Reported by Subject and/or Observed by Investigator.
Description: Safety and tolerability was measured by number of reported adverse events (serious and non-serious) and repeated clinical evaluation of physical examinations, vital signs, 12-lead electrocardiogram (ECG), 24-hour continuous cardiac monitoring, and laboratory tests (hematology/blood chemistry/urinalysis).
Time Frame: Screening (Day -5 for continuous cardiac monitoring) to Day 22
Population: All randomized patients who ingested at least one dose of study drug or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 4 | 9 | 8
participants
  Serious Adverse Events | 0 (0) | 0 (0) | 1 (0)
  Non-Serious Adverse Events | 0 (0) | 5 (0) | 5 (0)
  No Adverse Events Reported | 4 (0) | 4 (0) | 3 (0)

2. Primary Outcome: EVP-6124 Maximum Plasma Concentration (Cmax), Patients on Aripiprazole
Description: Blood samples for pharmacokinetic (PK) analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: All patients receiving aripiprazole.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 7 | 3
pg/mL
  Day 1 | 581.0 (149.8) | 210.0 (39.3)
  Day 21 | 2058.6 (393.2) | 968.3 (90.1)

3. Primary Outcome: EVP-6124 Time to Maximum Concentration (Tmax), Patients on Aripiprazole
Description: Blood samples for PK analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: All patients receiving aripiprazole.
Measure: Median (Full Range); unit: hr
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 7 | 3
hr
  Day 1 | 8.0 [2 to 8] | 8.0 [6 to 8]
  Day 21 | 6.0 [2 to 8] | 8.0 [1 to 8]

4. Primary Outcome: EVP-6124 Area Under the Curve (AUC[0-24 h]), Patients on Aripiprazole
Description: Blood samples for PK analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: All patients receiving aripiprazole.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 7 | 3
pg*hr/mL
  Day 1 | 10,966 (2831) | 3838 (1044)
  Day 21 | 42,042 (9623) | 20,560 (2699)

5. Primary Outcome: EVP-6124 Half-life (T[1/2]), Patients on Aripiprazole
Description: Blood samples for PK analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: Patients receiving aripiprazole for whom blood samples were available for analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 1 | 1
hr
  Day 1 | 39.0 (NA) — Data for only one patient were available. | 43.1 (NA) — Data for only one patient were available.
  Day 21 | NA (NA) — The patient withdrew consent after receiving study drug for 3 days. | 116.6 (NA) — Data for only one patient were available.

6. Primary Outcome: EVP-6124 Maximum Plasma Concentration (Cmax), Patients on Paliperidone/Risperidone
Description: Blood samples for PK analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: All patients receiving paliperidone/risperidone.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 1 | 5
pg/mL
  Day 1 | 315.0 (NA) — Data for only one patient were available. | 165.0 (40.2)
  Day 21 | 1510.0 (NA) — Data for only one patient were available. | 545.4 (130.2)

7. Primary Outcome: EVP-6124 Time to Maximum Concentration (Tmax), Patients on Paliperidone/Risperidone
Description: Blood samples for PK analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: All patients receiving paliperidone/risperidone.
Measure: Median (Full Range); unit: hr
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 1 | 5
hr
  Day 1 | 6.0 [NA to NA] — Data for only one patient were available. | 8.0 [6 to 8]
  Day 21 | 6.0 [NA to NA] — Data for only one patient were available. | 8.0 [8 to 8]

8. Primary Outcome: EVP-6124 Area Under the Curve (AUC[0-24 h]), Patients on Paliperidone/Risperidone
Description: Blood samples for PK analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: All patients receiving paliperidone/risperidone.
Measure: Mean (Standard Deviation); unit: pg*hr/ml
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 1 | 5
pg*hr/ml
  Day 1 | 6359 (NA) — Data for only one patient were available. | 3110 (852)
  Day 21 | 33,042 (NA) — Data for only one patient were available. | 11,888 (3095)

9. Primary Outcome: EVP-6124 Half-life (T[1/2]), Patients on Paliperidone/Risperidone
Description: Blood samples for PK analyses were taken before dosing with EVP-6124 on Days 1 and 21.
Time Frame: Days 1 and 21
Population: Patients receiving paliperidone/risperidone for whom blood samples were available for analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 1 | 2
hr
  Day 1 | 92.0 (NA) — Data for only one patient were available. | 45.8 (17.7)
  Day 21 | NA (NA) — Sample not analyzed. | 78.1 (8.3)

10. Secondary Outcome: N100 Gating Ratio
Description: N100 auditory evoked potential response (amplitude measured in microvolts) using the sensory gating paradigm. Measured by electroencephalography (EEG) as the amplitude ratio of test stimulus to conditioning stimulus. Plotted on a unitless scale of 0 to 2. Normalization is suggested by a lower value.
Time Frame: Days -1 to 20
Population: Subjects providing valid and measurable N100 responses.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 2 | 5 | 5
ratio | 1.648 (0.29) | 0.801 (0.19) | 0.951 (0.20)
Statistical Analysis 1: Comparison: Placebo vs EVP-6124 (1.0 mg/Day); Baseline value was the covariate and all values obtained during the treatment period were averaged together. This value was adjusted by regression against the baseline and estimation of a new value as if all subjects possessed the same baseline; Test type: Superiority or Other; p = 0.10, ANCOVA

11. Secondary Outcome: P50 Amplitude Difference
Description: P50 auditory evoked potential response (amplitude measured in microvolts) using sensory gating paradigm. Measured by EEG as amplitude difference (conditioning stimulus minus test stimulus). Plotted on a scale of -0.2 to 0.8 microvolts. Normalization is suggested by a higher value.
Time Frame: Days -1 to 20
Population: Subjects providing valid and measurable P50 responses.
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 2 | 5 | 5
microvolts | -0.17 (0.38) | 0.67 (0.21) | -0.06 (0.25)
Statistical Analysis 1: Comparison: Placebo vs EVP-6124 (1.0 mg/Day); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.07, ANCOVA

12. Secondary Outcome: MMN Summed Amplitude
Description: Mismatch negativity (MMN) auditory evoked potential response (amplitude in microvolts) using orienting paradigm. Measured by EEG and calculated as the voltage difference over 100-200 msec following stimulus onset (rare stimulus minus frequent stimulus). Plotted on a scale of -1.2 to 0.2 microvolts. Normalization is suggested by a more negative value.
Time Frame: Days -1 to 20
Population: Subjects providing valid and measurable MMN responses.
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 4 | 8 | 7
microvolts | 0.14 (0.33) | -1.15 (0.24) | -0.61 (0.25)
Statistical Analysis 1: Comparison: Placebo vs EVP-6124 (1.0 mg/Day) vs EVP-6124 (0.3 mg/Day); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.02, ANCOVA

13. Secondary Outcome: P300 Peak Amplitude
Description: P300 auditory evoked potential response (amplitude in microvolts) using orienting paradigm. Measured by EEG and calculated as the peak amplitude over 250-500 msec following stimulus onset (rare stimulus minus frequent stimulus). Plotted on a scale of -0.4 to 1.2 microvolts. Normalization is suggested by a more positive value.
Time Frame: Days -1 to 20
Population: Subjects providing valid and measurable P300 responses.
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Number analyzed (Participants) | 4 | 8 | 7
microvolts | -0.3 (0.31) | 1.08 (0.22) | 0.78 (0.24)
Statistical Analysis 1: Comparison: Placebo vs EVP-6124 (1.0 mg/Day) vs EVP-6124 (0.3 mg/Day); [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.008, ANCOVA

ADVERSE EVENTS:
Time Frame: Screening to Day 22
Arm/Group | Placebo | EVP-6124 (1.0 mg/Day) | EVP-6124 (0.3 mg/Day)
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9 | 1/8
Other Adverse Events (participants affected / at risk) | 0/4 | 5/9 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | EVP-6124 (1.0 mg/Day) (N=9) | EVP-6124 (0.3 mg/Day) (N=8)
Psychiatric symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | EVP-6124 (1.0 mg/Day) (N=9) | EVP-6124 (0.3 mg/Day) (N=8)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Psychiatric symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other